CLINICAL TRIAL: NCT02661750
Title: Safety and Efficacy of High Dose Bowel Preparation Solutions for Patients With Difficult To Clean Colons For Colonoscopy
Status: Completed | Type: Observational
Sponsor: Gastroenterology Services, Ltd. (Other)
Responsible Party: Sponsor
Other Study IDs: 2015-0004-02
Record Dates: First submitted 2016-01-19; First posted 2016-01-22 (Estimated); Last update posted 2021-07-27 (Actual); Status verified 2021-07

CONDITIONS: Preparation for Colonoscopy
Keywords: Cleansing the colon
MeSH Terms: interventions — Cathartics

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (5):
- Step 1: Patients who had inadequate preparations for colonoscopy with a standard dose of bowel cleansing agent.
  Interventions: Drug: Bowel Preparation
- Step 2: Patients who had inadequate preparations for colonoscopy with a step 1 dose of bowel cleansing agent.
  Interventions: Drug: Bowel Preparation
- Step 3: Patients who had inadequate preparations for colonoscopy with a step 2 dose of bowel cleansing agent.
  Interventions: Drug: Bowel Preparation
- Step 4: Patients who had inadequate preparations for colonoscopy with a step 3 dose of bowel cleansing agent.
  Interventions: Drug: Bowel Preparation
- Step 5: Patients who had inadequate preparations for colonoscopy with a step 4 dose of bowel cleansing agent.
  Interventions: Drug: Bowel Preparation

INTERVENTIONS:
Drug: Bowel Preparation — Standard 1/2 Dose: 153 g MiraLAX + 32 oz Gatorade 2 liters, 2 liters NuLYTELY, 1 liter MoviPrep, 16 oz (1 bottle) SuPREP, 10 oz (1 bottle) MagCitrate.
  Standard Full Dose: 306 g MiraLAX + 64 oz Gatorade, 4 liters NuLYTELY, 2 liters MoviPrep, 32 oz (2 bottles) SuPREP, 20 oz (2 bottles) MagCitrate.
  Step 1: 51 g MiraLAX* noon the day-prior; Full dose - 51 g MiraLAX 6 PM day-prior; 1/2 dose 4 hours before the colonoscopy.
  Step 2: 1/2 dose noon the day-prior; Full dose 6 PM the day-prior; 1/2 dose 4 hours before the colonoscopy.
  Step 3: Full dose noon the day-prior; Full dose 6 PM the day-prior; 1/2 dose 4 hours before the colonoscopy.
  Step 4: 1/2 dose 6 PM 2 days-prior; Full dose noon the day-prior; Full dose 6 PM the day-prior; 1/2 dose 4 hours before the colonoscopy.
  Step 5: Full dose 6 PM 2 days-prior; Full dose noon the day-prior; Full dose 6 PM the day-prior; 1/2 dose 4 hours before the colonoscopy.

SUMMARY:
The purpose of this study is to document the safety and effectiveness of high doses of liquids to clean the colon for colonoscopy in patients who had a previous colonoscopy with a poorly cleaned colon.

DETAILED DESCRIPTION:
Most of our patients use a standard dose of Gatorade (64 oz) and a tasteless laxative powder called MiraLAX (306 g) to clean their colons out for a colonoscopy. Occasionally, patients have chosen to use other FDA approved solutions to clean their colons including NuLYTELY, GoLytely, MoviPrep and SuPREP. Rarely patients choose to use high doses of MagCitrate.

Despite drinking all their liquid to clean their colon, a few patients have difficult to clean out colons and the quality of their colonoscopy preparation was not good. No one has ever studied what liquids to give these patients when they have another colonoscopy. Most doctors recommend using higher than standard doses of bowel cleaning liquids, but the safety and effectiveness of these higher doses has never been studied.

Patients will already have been assigned a higher than standard dose of a bowel cleaning liquid of their choice for their planned colonoscopy. This is our standard of care for cleaning out the colons of patients who previous had colonoscopies with colons that were not adequately cleaned. If the patient chooses to participate in this study, the plans to clean their colon will remain unchanged.

Before and during the study: The subject will clean out thier colon in the days before their colonoscopy just as they would have if they were not part of the study. They will be asked to fill out a short questionnaire before the colonoscopy about their experience with the liquid and the clean out process.

We would like to obtain a blood test (basic metabolic profile) that looks at each subject's kidney function within 3 months before their colonoscopy and before the IV is started for the colonoscopy. This involves a simple needle stick to draw 1 teaspoon (5 ml) of blood. If the subject had had blood tests done for other reasons within 3 months of their colonoscopy, these results can be used in place of the first blood sample.

The only research activity is the collection of patient's blood and the questionnaire the subject will fill out before the colonoscopy. The preparation to clean their colon and the actually colonoscopy will be unaffected by this research.

ELIGIBILITY:
Inclusion Criteria:

* Patients at least 18 years old planning to undergo an elective colonoscopy will be eligible for inclusion in our study if they had a previous colonoscopy with an inadequate preparation.

Exclusion Criteria:

* Patients who are pregnant.
* Patients with ileus, gastrointestinal obstruction, gastric retention, bowel perforation, toxic colitis or toxic megacolon would not be considered elective colonoscopies and are excluded.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients in our practice who are undergoing a routine colonoscopy who had an inadequate preparation for colonoscopy in the past
Sampling Method: Non-Probability Sample
Enrollment: 79 (Actual)
Dates: Start 2016-01 (Actual); Primary Completion 2021-01 (Actual); Study Completion 2021-01 (Actual)

PRIMARY OUTCOMES:
Bowel Cleanliness | at colonoscopy
  Measured by the Chicago Bowel Preparation Scale

SECONDARY OUTCOMES:
Bowel Cleanliness | at colonoscopy
  Measured by the Boston Bowel Preparation Scale
Bowel Cleanliness | at colonoscopy
  Measured by an adequate/inadequate bowel preparation scale
Patient tolerance | 1-2 days before colonoscopy measured at colonoscopy
  subject questionnaire
Electrolyte changes | at colonoscopy
  measured using a BMP before and after the colonoscopy preparation

CONTACTS AND LOCATIONS:
Locations (1):
- Gastroenterology Services, Downers Grove, Illinois, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Gerard DP, Gerard SF, Raiser MW. High-dose polyethylene glycol-3350 and gatorade solutions for patients with previous inadequate bowel preparations for colonoscopy are safe and effective. BMC Gastroenterol. 2023 May 11;23(1):146. doi: 10.1186/s12876-023-02663-0. PMID 37170191